CLINICAL TRIAL: NCT01452633
Title: Effect of Preincisional Local Analgesia on Post-Operative Pain in 10-12mm Lateral Port Sites
Brief Title: Study to Compare Reduction in Pain After Surgery With and Without Local Anesthesia During Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, James Droesch, Associate Professor, Obsterics/Gynecology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 241577-1
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Post Operative Pain
Keywords: pain; laparoscopy; reduction
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Preincision Placebo (Placebo Comparator): This group of patients will receive saline injection at study port site before incision
  Interventions: Drug: Saline will be injected at the study port site prior to incision
- Preincision Marcaine (Active Comparator): This group will receive marcaine injection at the study port site prior to incision
  Interventions: Drug: 0.25% bupivicaine will be injected at the study port site prior to incision
- Postincision Placebo (Placebo Comparator): This group of patients will receive preincisional marcaine and then saline injection at study port site prior to closure
  Interventions: Drug: 0.25% bupivicaine will be injected at the study port site prior to incision; Drug: Saline will be in injected into the port site prior to closure
- Postincision marcaine (Active Comparator): This group will receive preincisional marcaine and then marcaine injection at study port site prior to closure
  Interventions: Drug: 0.25% bupivicaine will be injected at the study port site prior to incision; Drug: 0.25% bupivicaine will be injected into the port site prior to closure

INTERVENTIONS:
Drug: 0.25% bupivicaine will be injected at the study port site prior to incision — Injection will precede the incision
  Other Names: marcaine
  Arms: Postincision Placebo; Postincision marcaine; Preincision Marcaine
Drug: Saline will be injected at the study port site prior to incision — Injection will precede incision
  Other Names: normal saline
  Arms: Preincision Placebo
Drug: Saline will be in injected into the port site prior to closure — Saline will be injected into the port site prior to the closure without any preincisional intervention
  Arms: Postincision Placebo
Drug: 0.25% bupivicaine will be injected into the port site prior to closure — 0.25% bupivicaine will be injected into the port site at closure without any preincisional intervention
  Other Names: marcaine
  Arms: Postincision marcaine

SUMMARY:
This study will help to answer the question, "Does injecting local anesthetic before laparoscopic instrument ports are placed decrease pain after surgery?" Patients participating will be randomly assigned to receive local anesthetic or saline injection at the site of a laparoscopic instrument port as part of their planned surgery. After surgery at 4 and 24 hours the patient will be asked to rate their pain on a simple chart.

DETAILED DESCRIPTION:
The literature is divided on the efficacy of preincisional local analgesia injections at laparoscopic port sites to decrease post operative pain. One reason for this lack of a clear conclusion is the fact that prior studies included small and large port sizes. Many small port sites have little pain associated with them so showing a reduction with medicine is statistically difficult. The investigators have noted that larger, lateral port sites which require fascial closure are the sites that patients consistently note pain at. Our protocol will include the use of 0.25% marcaine injections at all the surgical ports other than the large lateral port used for gynecologic laparoscopy. Patients would then be randomized and surgeons would be blinded as to which patients receive the marcaine or a saline injection at the large lateral port site. Visual analog pain scales will be assessed at 4 and 24 hours after surgery. An additional two arms have been added to include 50 patients randomized to 0.25% marcaine or saline injection just prior to incisional closure in the absence of any preincisional intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic surgery

Exclusion Criteria:

* Cardiovascular instability
* malignancies
* pulmonary conditions incompatible with laparoscopic surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in post-operative pain at large lateral port sites | 4 and 24 hours after surgery
  visual analog scoring of post-operative pain in a control and a treatment group

CONTACTS AND LOCATIONS:
Overall Officials: James N Droesch, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States